CLINICAL TRIAL: NCT00265616
Title: A Randomized Clinical Trial for the Treatment of Refractory Status Epilepticus
Brief Title: Treatment of Refractory Status Epilepticus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Andrea O. Rossetti, MD, Dr, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RSE study, protocol#62/06
Record Dates: First submitted 2005-12-13; First posted 2005-12-15 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Status Epilepticus
Keywords: Refractory status epilepticus,; coma-induction,; treatment,; propofol,; barbiturates,; efficacy,; safety.
MeSH Terms: conditions — Status Epilepticus | interventions — Propofol; Thiopental; Pentobarbital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): propofol, 2mg/kg as bolus, then titrated up to EEG burst-suppression as a continuous infusion; no maximum doses defined
  Interventions: Drug: propofol
- 2 (Active Comparator): thiopental/pentobarbital, 2mg/kg as bolus, then titrated up to EEG burst-suppression as a continuous infusion; no maximum doses defined
  Interventions: Drug: thiopental/pentobarbital

INTERVENTIONS:
Drug: propofol — liquid, mg/kg.h, titrated after EEG
  Other Names: Disoprivan
  Arms: 1
Drug: thiopental/pentobarbital — liquid, mg/kg.h, titrated after EEG
  Other Names: Pentotal /Thiopentone
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether propofol or barbiturates should be preferred in the treatment of status epilepticus (continuous seizure activity) refractory to 2 standard antiepileptic agents.

DETAILED DESCRIPTION:
Refractory status epilepticus (SE) develops in 31%-44% of patients with SE, with a mortality of 16%-23%. Coma induction is advocated for its management. Propofol and barbiturates are the most used agents, but no comparative study has been performed. In consideration of the uncertainty regarding the relative effectiveness, despite several retrospective data, a prospective investigation is needed.

The objective is to assess the effectiveness (SE control, adverse events) of a first course of propofol versus barbiturates in the treatment of refractory SE, in adults with refractory SE not due to cerebral anoxia.

Comparison: Coma induction with standardized doses of propofol or barbiturates titrated towards burst-suppression on EEG, then assessment of the proportion of patients achieving a control of SE.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory status epilepticus not due to cerebral anoxia, needing coma induction for clinical management.

Exclusion Criteria:

* Age < 16 years old.
* Known pregnancy.
* Cerebral anoxia as SE etiology.
* Epilepsia partialis continua (simple partial SE).
* Known intolerance to the study drugs.
* Known mitochondrial disorder, hyperlipidemia, or significant rhabdomyolysis.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea O. Rossetti, MD, Principal Investigator — BrighamHospital/CHUV
Locations (5):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
- Switzerland (3):
  - Inselspital, Bern, Canton of Bern
  - CHUV, Lausanne, Canton of Vaud
  - Hôpitaux Universitaires de Genève, Geneva

REFERENCES:
- [Result] Rossetti AO, Milligan TA, Vulliemoz S, Michaelides C, Bertschi M, Lee JW. A randomized trial for the treatment of refractory status epilepticus. Neurocrit Care. 2011 Feb;14(1):4-10. doi: 10.1007/s12028-010-9445-z. PMID 20878265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Rcruitment in participating centers took part between 2006 and 2010.
Groups:
- Propofol: titrated to electroencephalographic burst-suppression (intravenous load as per protocol, then following the EEG);no maximum doses defined.
- Thiopental/Pentobarbital: titrated to electroencephalographic burst-suppression (intravenous load as per protocol, then following the EEG); no maximum doses defined.
Period: Overall Study
Arm/Group | Propofol | Thiopental/Pentobarbital
Started | 14 | 9
Completed | 14 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol; Thiopental/Pentobarbital: titrated to electroencephalographic burst-suppression (intravenous load as per protocol, then following the EEG)
- Total: Total of all reporting groups
Arm/Group | Propofol | Thiopental/Pentobarbital | Total
Number analyzed (Participants) | 14 | 9 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 9 | 4 | 13
  >=65 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 7 | 3 | 10
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 7
  Switzerland | 9 | 7 | 16

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Outcome at Day 21
Description: Return to baseline clinical conditions (i.e.: no new handicap, no death)
Time Frame: 21 days
Measure: Number; unit: participants
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
participants | 5 | 3
Statistical Analysis 1: Comparison: Propofol vs Thiopental/Pentobarbital; Test type: Superiority or Other; p = 1.00, Fisher Exact

2. Secondary Outcome: Patients With Infectious Complications Requiring Specific Treatment
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
participants | 7 | 6
Statistical Analysis 1: Comparison: Propofol vs Thiopental/Pentobarbital; Test type: Superiority or Other; p = 0.67, Fisher Exact

3. Secondary Outcome: Patients With Hypotension Requiring Specific Treatment
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
participants | 7 | 5
Statistical Analysis 1: Comparison: Propofol vs Thiopental/Pentobarbital; Test type: Superiority or Other; p = 1.00, Fisher Exact

4. Secondary Outcome: Patients With Propofol Infusion Syndrome
Description: Propofol infusion syndrome (PRIS) is a severe metabolic alteration with elevation of lactate, CK, and triglycerides.
Time Frame: 10 days
Measure: Number; unit: participants
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
participants | 1 | 0

5. Primary Outcome: Refractory Status Epilepticus Controlled With First Course of Study Drug
Description: Control of status epilepticus refractory to benzodiazepines and a first antiepileptic drug after administration of the study drug; dichotomous assessment (yes/no)
Time Frame: after return of continuous EEG activity (typically after 36 hours - 5 days)
Population: Number of patients fulfilling primary outcome criteria
Measure: Number; unit: participants
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
participants | 6 | 2
Statistical Analysis 1: Comparison: Propofol vs Thiopental/Pentobarbital; Test type: Superiority or Other; p = 0.4, Fisher Exact

6. Secondary Outcome: Intubation Time in Survivors
Time Frame: Up to 3 months
Measure: Median (Full Range); unit: days
Arm/Group | Propofol | Thiopental/Pentobarbital
Number analyzed (Participants) | 14 | 9
days | 4 [2 to 28] | 13.5 [8 to 70]
Statistical Analysis 1: Comparison: Propofol vs Thiopental/Pentobarbital; Test type: Superiority or Other; p = 0.03, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Propofol | Thiopental/Pentobarbital
Serious Adverse Events (participants affected / at risk) | 1/14 | 1/9
Other Adverse Events (participants affected / at risk) | 0/14 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol (N=14) | Thiopental/Pentobarbital (N=9)
propofol infusion syndrome (non fatal) (Cardiac disorders) | 1 (1) | 0 (0)
paralytic ileus (fatal) (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No